CLINICAL TRIAL: NCT02141152
Title: Next pErsonalized Cancer tX With mulTi-omics and Preclinical Model: The Master Protocol
Brief Title: Next pErsonalized Cancer tX With mulTi-omics and Preclinical Model
Acronym: NEXT-1
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD,PhD, Samsung Medical Center
Other Study IDs: 2013-10-017
Record Dates: First submitted 2014-02-10; First posted 2014-05-19 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fresh tissue or FFPE
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- gastric cancer: This study will recruit a total of 130 gastric cancer patients. It is expected to recruit about 250 gastric cancer patients per year. Since the incidence of each mutation is low, the different types of mutations are assumed to be mutually exclusive. So, about 30% of these patients are expected to have a mutation with a target drug. Overall response (OR) is the primary endpoint of this study. OR rate (ORR) will be compared between the group (called targeted group) of patients who have a mutation with a target drug and that (called untargeted group) of patients who have no mutation. The ORR is expected to be about 25% for the targeted group and about 5% for the untargeted group. With N=130 gastric cancer patients, about 39 patients will belong to the targeted group and about 91 will belong to the untargeted group. The chi-square test with a 2-sided alpha=5% has 89% of power. The study on gastric cancer will take 7 months for patient accrual.
- colorectal cancer: This study will recruit a total of 130 colorectal cancer patients. It is expected to recruit about 300 colorectal cancer patients per year. About 25% of these patients are expected to have a mutation with a target drug. ORR will be compared between the targeted group and the untargeted group. The median ORR is expected to be about 25% for the targeted group and about 5% for the untargeted group. With N=130 colorectal cancer patients, about 33 patients will belong to the targeted group and about 97 will belong to the untargeted group. The chi-square test with a 2-sided alpha=5% has 87% of power. The study on colorectal cancer will take about 6 months for accrual.
- biliary tract cancer/pancreatic cancer: This study will recruit a total of 78 biliary tract cancer/pancreatic cancer patients. It is expected to recruit about 100 biliary tract cancer/pancreatic cancer patients per year. About 20% of these patients are expected to have a mutation with a target drug. ORR will be compared between the targeted group and the untargeted group. The ORR is expected to be about 35% for the targeted group and about 5% for the untargeted group. With N=78 biliary tract cancer/pancreatic cancer patients, about 16 patients will belong to the targeted group and about 62 will belong to the untargeted group. The chi-square test with a 2-sided alpha=5% has 87% of power. The study on biliary tract cancer/pancreatic cancer will take about 7 months for accrual.
- Rare cancer: Rare cancer is hepatocellular carcinoma, melanoma and neuroendocrine tumor. This study will recruit a total of 87 hepatocellular carcinoma/rare cancer patients. It is expected to recruit about 150 biliary tract cancer/pancreatic cancer patients per year. About 25% of these patients are expected to have a mutation with a target drug. ORR will be compared between the targeted group and the untargeted group. The ORR is expected to be about 30% for the targeted group and about 5% for the untargeted group. With N=87 biliary tract cancer/pancreatic cancer patients, about 22 patients will belong to the targeted group and about 65 will belong to the untargeted group. The chi-square test with a 2-sided alpha=5% has 86% of power. The study on biliary tract cancer/pancreatic cancer will take about 7 months for accrual.
- genitourinary cancer

SUMMARY:
The next generation of personalized medical treatment according to the type of personal genetic information are evolving rapidly. The genome analysis needs systematic infra and database based on personal genetic information Therefore, a big data of genome-clinical information is important.

To determine the feasibility of the use of tumor's molecular profiling and targeted therapies in the treatment of advanced cancer and to determine the clinical outcome(PFS, duration of response and overall survival) of patients with advanced cancer, the investigators are going to take a fresh tissue of patients and process molecular profiling and receive molecular profile directed treatments.

DETAILED DESCRIPTION:
This study nickname is NEXT-1 trial(Next pErsonalized cancer tX with mulTi). A single-center, open label trial to analysis of genetic information in advanced cancer.

If the target is to be confirmed by molecular profile, the subgroup is going to Umbrella trial type.

defined below: NEXT 1 trial is screening and feasibility -> NEXT trial is BASKET/umbrella study screening protocol(Molecular screening prolongs survival)->NEXT-1.1(gastric cancer),NEXT-1.2(colorectal cancer),NEXT-1.3(biliary tract cancer/pancreatic cancer),NEXT-1.4(Rare cancer),NEXT-1.5(genitourinary cancer)

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed metastatic malignancy
* Written informed consent

Exclusion Criteria:

* patients who do not agree with biopsy
* patients who do not have enough tissue for acquisition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with treatment-refractory malignancy
Sampling Method: Probability Sample
Enrollment: 895 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Response rate | expected average of 3 years
  To compare response rate (RR) (per RECIST 1.1) in patient cohort with molecularly matched treatment (in practice or in the context of clinical trials) versus RR in patient cohort with non-matched treatment based on molecular profiling

SECONDARY OUTCOMES:
Progression Free Survival | expected average of 3 years
  To compare PFS in patient cohort with molecularly matched treatment (in practice or in the context of clinical trials) versus PFS in patient cohort with non-matched treatment based on molecular profiling
feasibility | expected average of 3 years
  To evaluate changes in the tumor's molecular profile on serial biopsies
feasibility | expected average of 3 years
  To establish n of 1 preclinical model for each patient whenever feasible

CONTACTS AND LOCATIONS:
Overall Officials: Won Ki Kang, MD, Study Chair — Division of Hematology-Oncology, Department of Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim ST, Kim KM, Kim NKD, Park JO, Ahn S, Yun JW, Kim KT, Park SH, Park PJ, Kim HC, Sohn TS, Choi DI, Cho JH, Heo JS, Kwon W, Lee H, Min BH, Hong SN, Park YS, Lim HY, Kang WK, Park WY, Lee J. Clinical Application of Targeted Deep Sequencing in Solid-Cancer Patients and Utility for Biomarker-Selected Clinical Trials. Oncologist. 2017 Oct;22(10):1169-1177. doi: 10.1634/theoncologist.2017-0020. Epub 2017 Jul 12. PMID 28701572